CLINICAL TRIAL: NCT06204146
Title: The Effect of Massage Applied to Preterm Infants On Growth and Stress
Brief Title: The Effect of Massage on Growth And Stress And Stress ,Department of Nursing,
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EMİNE SARIKAMIŞ KALE (Other)
Responsible Party: Sponsor-Investigator, EMİNE SARIKAMIŞ KALE, Phd student, Hasan Kalyoncu University
Organization: Hasan Kalyoncu University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017/015
Record Dates: First submitted 2023-10-24; First posted 2024-01-12 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Preterm
Keywords: preterm
MeSH Terms: conditions — Premature Birth | interventions — Massage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- massage (Experimental): massage was applied to the infants in the experimental group three times daily for 10 days,
  Interventions: Behavioral: massage
- control (No Intervention): the control group received the usual care

INTERVENTIONS:
Behavioral: massage — stressn level and preterm growth
  Arms: massage

SUMMARY:
The aim of this thesis is to exprementally investigate the effect of massage applied to preterm infants on growth and stress. While the population of the research is preterm infants at the neonatal intensive care unit of a Medicalpark Batman Hospital between January 2018 and February 2019, the sample is 60 preterm infants suitable for inclusion criteria. Research data was collected using Preterm Infant Information Form, Preterm Follow-up Form and Newborn Stress Scale. While massage was applied to the infants in the experimental group three times daily for 10 days, the control group received the usual care. Weight, length and head circumference of infants in both experimental and control group were measured by the researcher on 1., 5. and 10. days. In order to evaluate stess level of the massage applied infants, camera records of the infants were taken 15 minutes before and after the massage on 1., 5. and 10. days. Camera records of the infants in the control group were also taken at the same time with those in the experimental group. Camera records were watched and stress level of the infants were evaluated by two observers blind to the research. The data analyses were carried out using In-class Correlation, Frequency, Levene, Two-Way ANOVA for Mixed Measured, Repeated ANOVA tests

DETAILED DESCRIPTION:
The aim of this thesis is to exprementally investigate the effect of massage applied to preterm infants on growth and stress

ELIGIBILITY:
Inclusion Criteria:

- Gestational age at birth below 36 weeks + 6 days, Body weight over 1000 g, Do not have any diseases or congenital disorders, Babies who are allowed to be massaged by the NICU's neonatologist was determined as .

Exclusion Criteria:

-

Ages: 27 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2019-06-07 (Actual); Study Completion 2019-07-10 (Actual)

PRIMARY OUTCOMES:
Weight | 10 days
  physiological parameter is analyzed, it is observed first day and ten day the baby weight
length | 10 days
  physiological is analyzed, it is observed first day and ten day the baby length
head circumference | 10 days
  physiological parameter is analyzed, it is observed first day and ten day the baby head circumference
newborn stres scale | 10 days
  it is an assessment tool developed to evaluate the stress level of newborn. 0-2 point each item min max 16point each subscale

CONTACTS AND LOCATIONS:
Overall Officials: emine sarıkamış kale, MSc, Principal Investigator — Hasan Kalyoncu University
Locations (1):
- Emine Sarıkamış Kale, Batman, Merkez, Turkey (Türkiye)